CLINICAL TRIAL: NCT00454116
Title: A Phase II, Double Blind, Placebo Controlled, Randomised Study to Assess the Efficacy and Safety of 2 Doses of ZACTIMA™(ZD6474) in Combination With FOLFIRI vs FOLFIRI Alone for the Treatment of Colorectal Cancer in Patients Who Have Failed Therapy With an Oxaliplatin and Fluoropyrimidine Containing Regimen
Brief Title: A Phase II, Double Blind Study of 2 Doses of ZACTIMA™(ZD6474) in Combination With FOLFIRI vs FOLFIRI Alone for the Treatment of Colorectal Cancer in Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4200C00048; 2006-005023-42 (EudraCT Number)
Record Dates: First submitted 2007-03-28; First posted 2007-03-30 (Estimated); Results first posted 2011-05-24 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Cancer
Keywords: Colon Cancer; Rectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — vandetanib; IFL protocol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): FOLFIRI + placebo vandetanib
  Interventions: Drug: FOLFIRI
- 2 (Experimental): FOLFIRI + low dose vandetanib
  Interventions: Drug: Vandetanib; Drug: FOLFIRI
- 3 (Experimental): FOLFIRI + high dose vandetanib
  Interventions: Drug: Vandetanib; Drug: FOLFIRI

INTERVENTIONS:
Drug: Vandetanib — once daily oral tablet two doses
  Other Names: ZD6474; ZACTIMA™
  Arms: 2; 3
Drug: FOLFIRI — Intravenous infusion

SUMMARY:
The purpose of this study is to assess the efficacy and safety of 2 doses of ZACTIMA™ (ZD6474) in combination with FOLFIRI vs FOLFIRI alone for the treatment of colorectal cancer in patients who have failed therapy with an oxaliplatin and fluoropyrimidine containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal cancer
* Have failed therapy with an oxaliplatin and fluoropyrimidine containing regimen defined as:
* Progression on or following treatment for metastatic colorectal cancer
* Progression within 12 months of adjuvant chemotherapy for colorectal cancer

Exclusion Criteria:

* Previous treatment with small molecule tyrosine kinase inhibitors of VEGFR or EGFR eg, erlotinib, gefitinib. Prior monoclonal antibodies are permitted, eg, cetuximab, bevacizumab.
* Previous adjuvant therapy with irinotecan within 12 months of randomization
* More than one prior course of chemotherapy for treatment of metastatic colorectal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (21):
- United States (4):
  - Research Site, Ann Arbor, Michigan
  - Research Site, New York, New York
  - Research Site, Nashville, Tennessee
  - Research Site, Salt Lake City, Utah
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, Ramos Mejía
  - Research Site, Rosario
  - Research Site, Santa Fe
  - Research Site, Vicente López
- Norway (3):
  - Research Site, Bergen
  - Research Site, Oslo
  - Research Site, Stavanger
- Research Site, Seoul, South Korea
- Spain (4):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Jaén
  - Research Site, Lleida
- United Kingdom (4):
  - Research site, Belfast, Northern Ireland
  - Research Site, Aberdeen
  - Research Site, Leicester
  - Research Site, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient randomised 14 March 2007, last patient randomised 21 Jan 2008, data cut off data 31 March 2008
Groups:
- Vandetanib 100 mg Plus FOLFIRI: vandetanib 100 mg plus FOLFIRI
- Vandetanib 300 mg Plus FOLFIRI: vandetanib 300 mg plus FOLFIRI
- Placebo Plus FOLFIRI: placebo plus FOLFIRI
Period: Overall Study
Arm/Group | Vandetanib 100 mg Plus FOLFIRI | Vandetanib 300 mg Plus FOLFIRI | Placebo Plus FOLFIRI
Started | 35 (randomised patients) | 36 (randomised patients) | 35 (randomised patients)
Completed | 8 (ongoing study treatment at data cut-off) | 7 (ongoing study treatment at data cut-off) | 7 (ongoing study treatment at data cut-off)
Not Completed | 27 | 29 | 28
Not completed — Adverse Event | 5 | 11 | 9
Not completed — Condition under investigation worsened | 17 | 13 | 18
Not completed — Withdrawal by Subject | 3 | 3 | 1
Not completed — Other | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vandetanib 100 mg Plus FOLFIRI | Vandetanib 300 mg Plus FOLFIRI | Placebo Plus FOLFIRI | Total
Number analyzed (Participants) | 35 | 36 | 35 | 106
Age, Continuous [Mean (Full Range); unit: years] | 57 [39 to 80] | 57 [30 to 73] | 59 [37 to 73] | 58 [30 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 15 | 43
  Male | 20 | 23 | 20 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With an Objective Disease Progression Event
Description: Number of patients with objective disease progression or death (by any cause in the absence of objective progression)
Time Frame: Tumour assessments carried out at screening and then as per site clinical practice until objective progression. The only additional mandatory tumour assessment visit is at the point of data cut-off (28 March 2008 +/-3 days)
Measure: Number; unit: Participants
Arm/Group | Vandetanib 100 mg Plus FOLFIRI | Vandetanib 300 mg Plus FOLFIRI | Placebo Plus FOLFIRI
Number analyzed (Participants) | 35 | 36 | 35
Participants | 20 | 24 | 24

ADVERSE EVENTS:
Arm/Group | Vandetanib 100 mg Plus FOLFIRI | Vandetanib 300 mg Plus FOLFIRI | Placebo Plus FOLFIRI
Serious Adverse Events (participants affected / at risk) | 8/35 | 13/36 | 12/35
Other Adverse Events (participants affected / at risk) | 32/35 | 36/36 | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib 100 mg Plus FOLFIRI (N=35) | Vandetanib 300 mg Plus FOLFIRI (N=36) | Placebo Plus FOLFIRI (N=35)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 2 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 2
ANGINA PECTORIS (Cardiac disorders) | 1 | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 3 | 2
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 2
ILEUS (Gastrointestinal disorders) | 1 | 0 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1
PROCTITIS (Gastrointestinal disorders) | 1 | 0 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
PYREXIA (General disorders) | 1 | 3 | 3
CHEST PAIN (General disorders) | 1 | 0 | 0
CENTRAL LINE INFECTION (Infections and infestations) | 1 | 2 | 0
BETA HAEMOLYTIC STREPTOCOCCAL INFECTION (Infections and infestations) | 0 | 1 | 0
CELLULITIS (Infections and infestations) | 1 | 0 | 0
EPSTEIN-BARR VIRUS INFECTION (Infections and infestations) | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 1 | 1
SEPSIS (Infections and infestations) | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
VIRAL INFECTION (Infections and infestations) | 0 | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib 100 mg Plus FOLFIRI (N=35) | Vandetanib 300 mg Plus FOLFIRI (N=36) | Placebo Plus FOLFIRI (N=35)
NEUTROPENIA (Blood and lymphatic system disorders) | 16 | 17 | 19
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 6 | 3
LEUKOPENIA (Blood and lymphatic system disorders) | 2 | 2 | 4
ANAEMIA (Blood and lymphatic system disorders) | 1 | 2 | 3
DIARRHOEA (Gastrointestinal disorders) | 18 | 26 | 17
NAUSEA (Gastrointestinal disorders) | 17 | 12 | 18
STOMATITIS (Gastrointestinal disorders) | 10 | 15 | 16
VOMITING (Gastrointestinal disorders) | 9 | 6 | 12
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 | 4 | 8
CONSTIPATION (Gastrointestinal disorders) | 7 | 6 | 7
DYSPEPSIA (Gastrointestinal disorders) | 4 | 6 | 6
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 1 | 3
FLATULENCE (Gastrointestinal disorders) | 3 | 1 | 0
ORAL PAIN (Gastrointestinal disorders) | 3 | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 2 | 1
DRY MOUTH (Gastrointestinal disorders) | 0 | 1 | 2
HAEMORRHOIDS (Gastrointestinal disorders) | 2 | 0 | 1
PROCTALGIA (Gastrointestinal disorders) | 2 | 1 | 0
FATIGUE (General disorders) | 10 | 9 | 9
ASTHENIA (General disorders) | 7 | 6 | 6
PYREXIA (General disorders) | 6 | 3 | 3
OEDEMA PERIPHERAL (General disorders) | 1 | 3 | 3
CHILLS (General disorders) | 1 | 1 | 2
INJECTION SITE REACTION (General disorders) | 2 | 0 | 1
CENTRAL LINE INFECTION (Infections and infestations) | 0 | 4 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 4 | 0
NASOPHARYNGITIS (Infections and infestations) | 3 | 1 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 3 | 2
ELECTROCARDIOGRAM QT PROLONGED (Infections and infestations) | 4 | 8 | 1
ANOREXIA (Metabolism and nutrition disorders) | 11 | 10 | 15
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 1 | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 3 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
LETHARGY (Nervous system disorders) | 5 | 2 | 4
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 | 2 | 5
DIZZINESS (Nervous system disorders) | 2 | 4 | 4
HEADACHE (Nervous system disorders) | 2 | 3 | 1
CHOLINERGIC SYNDROME (Nervous system disorders) | 0 | 2 | 1
DYSGEUSIA (Nervous system disorders) | 2 | 2 | 2
INSOMNIA (Psychiatric disorders) | 5 | 2 | 0
ANXIETY (Psychiatric disorders) | 0 | 3 | 2
HAEMATURIA (Renal and urinary disorders) | 0 | 3 | 0
DYSURIA (Renal and urinary disorders) | 0 | 2 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 8 | 22 | 6
ALOPECIA (Skin and subcutaneous tissue disorders) | 12 | 10 | 15
PRURITUS (Skin and subcutaneous tissue disorders) | 2 | 5 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 4 | 2
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
ACNE (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
HYPERTENSION (Vascular disorders) | 0 | 4 | 2
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 0 | 2 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 2
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 2
LACRIMATION INCREASED (Eye disorders) | 2 | 0 | 1
VISION BLURRED (Eye disorders) | 0 | 1 | 2
SKIN INFECTION (Infections and infestations) | 0 | 2 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.